CLINICAL TRIAL: NCT01205568
Title: Safety and Efficacy of the Cutting Balloon to Treat Resistant Pulmonary Artery Stenosis
Brief Title: Cutting Balloon Study
Acronym: CB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Kathy Jenkins, Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0502027R; 75593
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Artery Stenosis
MeSH Terms: conditions — Stenosis, Pulmonary Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Resistant Pulmonary Artery Stenosis (Experimental): Vessels with resistant PA stenosis were identified during catheterization and eligible vessels were randomized to Cutting Balloon or High Pressure Balloon Dilation
  Interventions: Device: Transcatheter Cutting Balloon therapy; Procedure: High Pressure Balloon Angioplasty

INTERVENTIONS:
Device: Transcatheter Cutting Balloon therapy
Procedure: High Pressure Balloon Angioplasty

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of transcatheter Cutting Balloon therapy for branch pulmonary artery stenosis resistant to low pressure dilation.

DETAILED DESCRIPTION:
The proposed study will be a prospective, multi-center, randomized, blinded trial comparing 2 treatments for pulmonary artery stenosis. Specifically, vessels that fail to respond to balloon inflation at 8 ATM will be individually randomized to 1 of 2 treatment pathways. In the first treatment pathway, the vessel is dilated using a CB, followed by additional low pressure balloon dilation (< 8ATM). In the second pathway,the vessel is dilated with high pressure balloon angioplasty, with balloon inflation pressures exceeding 15 ATM. Cross-over therapy will be permitted for failed high pressure treatment starting with enrollment of patient #15. The primary outcome assessment for efficacy will be a comparison of percent change in minimum lumen diameter before and after randomized therapy, as determined by a core laboratory blinded to pathway assignment. The primary outcome assessment for safety will be a comparison of the proportion of vessel dilations resulting in any serious adverse events, as determined by the Data and Safety Monitoring Board. Patient-level safety endpoints will also be tabulated. Patients can have multiple vessels enrolled; analytical techniques will adjust for potential intra-patient correlation.

ELIGIBILITY:
Inclusion Criteria:

Patient Inclusion Criteria (Determined Prior to Cardiac Catheterization)

a. At least 1 branch pulmonary artery stenosis referred for planned catheterization for PA dilation b. At least one of the following: i.greater than one half systemic right ventricular pressure ii. regional decrease in pulmonary blood flow by lung scan iii. elevated pulmonary artery pressures (> 20 mmHg MPAP) iv. cyanosis at least in part due to PA stenosis c. Informed consent of patient and/or parent/guardian; assent of mature minors d. Agreement to participate in protocol, including follow-up testing

Vessel Inclusion Criteria (Determined During Cardiac Catheterization)

1. Native pulmonary artery or branch which fails balloon dilation up to 8 ATM; as defined by failure to eliminate a waist
2. Native pulmonary artery or branch with a balloon waist diameter less than 7.5 mm (i.e.,0.5 mm less than the largest available CB) with dilation at 8 ATM
3. All eligible vessels that are dilated during the catheterization must be enrolled as study vessels; "off-study" use of Cutting Balloons or high pressure dilations in eligible vessels is not allowed.

Exclusion Criteria:

3. Patient Exclusion Criteria (Determined Prior to Cardiac Catheterization)

1. Prior pulmonary artery angioplasty or surgery on the vessel within the previous 6 weeks
2. Pregnancy

Vessel Exclusion Criteria (Determined During Cardiac Catheterization)

1. Vessel with an aneurysm from a prior dilation or surgery, defined as a local enlargement of the vessel greater than 100% of the lumen diameter both proximally and distally to the aneurysm. The maximum aneurysm diameter and vessel lumen diameter proximal and distal to the aneurysm will be recorded. The location of the aneurysm relative to the angioplasty site will be determined and reported as proximal, distal, or in the region of waist formation.
2. Prior stent placement associated with the obstruction

i. balloon inflation for the purpose of expanding the diameter of the stent along its length with no residual waist proximal or distal to the stent edges ii. balloon inflation resulting in waist formation within the edges of a stent iii. dilation of a vessel through the cells of a stent c. Unifocalized nor non-unifocalized systemic to pulmonary artery collaterals. d. A vessel requiring therapy at a site not amenable to delivery or safe positioning of a Cutting Balloon device due to unfavorable anatomy as determined by the physician and based on as assessment of vessel angles, size, length, and proximity to other vessels.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2003-08-01 (Actual); Primary Completion 2009-03-17 (Actual); Study Completion 2009-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Jenkins, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (6):
- United States (6):
  - University of California at San Francisco, San Francisco, California
  - Children's Hospital Boston, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital, Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among 73 patients, 331 stenotic vessels were identified. 86 vessels were not eligible and 245 vessels were potentially eligible. 72 vessels were considered successfully treated after low-pressure dilation. 173 met eligibility. 66 vessels were randomized to High Pressure Balloon (HPB) and 107 vessels were randomized to Cutting Balloon (CB).
Units Other Than Participants: Vessels
Groups:
- Cutting Balloon (CB): Resistant Vessels with Pulmonary Artery Stenosis were identified during catheterization and vessels were randomized to Cutting Balloon dilation.
- High Pressure Balloon (HPB): Resistant Vessels with Pulmonary Artery Stenosis were identified during catheterization and vessels were randomized to High Pressure Balloon dilation.
Period: Overall Study
Arm/Group | Cutting Balloon (CB) | High Pressure Balloon (HPB)
Started | 65; 107 Vessels (26 patients received only CB therapy, 39 patients received both CB and HPB therapy.) | 47; 66 Vessels (8 patients received only HPB therapy, 39 patients received both CB and HPB therapy.)
Completed | 65; 106 Vessels | 47; 65 Vessels
Not Completed | 0; 1 Vessels | 0; 1 Vessels

BASELINE CHARACTERISTICS:
Population: Baseline data prior to vessel randomization
Units Other Than Participants: Vessels
Groups:
- Patients With Resistant Pulmonary Artery Stenosis: Vessels with resistant PA stenosis were identified during catheterization and eligible vessels were randomized to Cutting Balloon or High Pressure Balloon Dilation.
  171 vessels in 73 patients were studied. Individual participants could have vessels randomized to one or both arms of the trial.
Arm/Group | Patients With Resistant Pulmonary Artery Stenosis
Number analyzed (Participants) | 73
Number analyzed (Vessels) | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 72
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 73
Greater than 1/2 systemic RV pressure [Count of Participants; unit: Participants] | 60
Regional decrease in pulmonary flow [Count of Participants; unit: Participants] | 58
Elevated PA pressure (mean >20) [Count of Participants; unit: Participants] | 47
Cyanosis in part due to PA stenosis [Count of Participants; unit: Participants] | 19

OUTCOME MEASURES:

1. Primary Outcome: Acute Change in Minimum Lumen Diameter Immediately Post-intervention
Description: The primary efficacy outcome is the percent change in minimum lumen diameter from pre-intervention to immediately post-intervention as measured by angiography.
Time Frame: Pre-intervention to immediate post-intervention (approximately 10 minutes)
Population: Vessels with resistant Pulmonary Artery Stenosis were identified during catheterization and eligible vessels were randomized to Cutting Balloon or High Pressure Balloon Dilation. Patients had variable number of eligible vessels. Each eligible vessel was randomized at the time of procedure.
Measure: Mean (Standard Deviation); unit: percentage change
Units Other Than Participants: vessels
Groups:
- Patients With Resistant Pulmonary Artery Stenosis: Vessels with resistant Pulmonary Artery Stenosis were identified during catheterization and eligible vessels were randomized to Cutting Balloon or High Pressure Balloon Dilation.
Arm/Group | Patients With Resistant Pulmonary Artery Stenosis
Number analyzed (Participants) | 73
Number analyzed (vessels) | 171
percentage change
  Cutting Balloon: number analyzed (Participants) | 65
  Cutting Balloon: number analyzed (vessels) | 106
  Cutting Balloon | 85.1 (77.1)
  High Pressure Balloon Dilation: number analyzed (Participants) | 47
  High Pressure Balloon Dilation: number analyzed (vessels) | 65
  High Pressure Balloon Dilation | 52.4 (66)

2. Secondary Outcome: Percent Change in Minimum Lumen Diameter at 3 Months Post-intervention
Description: Late percent change in minimum lumen diameter from pre-intervention to follow-up angiography.
Time Frame: 3 months post-intervention
Population: Vessels with resistant Pulmonary Artery Stenosis were identified during catheterization and eligible vessels were randomized to Cutting Balloon or High Pressure Balloon Dilation.
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: vessels
Arm/Group | Patients With Resistant Pulmonary Artery Stenosis
Number analyzed (Participants) | 26
Number analyzed (vessels) | 76
percent change
  Cutting Balloon: number analyzed (Participants) | 25
  Cutting Balloon: number analyzed (vessels) | 45
  Cutting Balloon | 75.6 (97.8)
  High Pressure Balloon Dilation: number analyzed (Participants) | 21
  High Pressure Balloon Dilation: number analyzed (vessels) | 31
  High Pressure Balloon Dilation | 42.2 (66.9)

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events from the time of enrollment to follow-up assessment 2-4 months after the intervention.
Groups:
- Patients With Resistant Pulmonary Artery Stenosis: Vessels with resistant Pulmonary Artery Stenosis were identified during catheterization and eligible vessels were randomized to Cutting Balloon (CB) or High Pressure Balloon Dilation (HPB). Of the 73 patients, 26 received CB dilation only, 8 patients received HPB dilation only, and 39 patients received both CB and HPB dilations. Therefore, 65/73 patients were exposed to CB and 47/73 patients were exposed to HPB. Due to the overlap in treatment amongst patients, adverse events are reported on the patient level and not by intervention type.
Arm/Group | Patients With Resistant Pulmonary Artery Stenosis
Serious Adverse Events (participants affected / at risk) | 0/73
Other Adverse Events (participants affected / at risk) | 16/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Resistant Pulmonary Artery Stenosis (N=73)
Device malfunction (Cardiac disorders) | 2 (2)
Balloon Rupture (Cardiac disorders) | 3 (3)
Balloon caught on stent (Cardiac disorders) | 1 (1)
Fracture of catheter shaft (Cardiac disorders) | 1 (1)
Pulmonary Edema (Cardiac disorders) | 10 (10)
Intravascular tear (Cardiac disorders) | 1 (1)
Hemoptysis, hypotension (Cardiac disorders) | 1 (1)
Heart Block (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No